CLINICAL TRIAL: NCT01559909
Title: Effect of Brim Height Using Vacuum Assisted Technology With Transfemoral Amputees
Brief Title: Effect of Socket Wall Height With Vacuum Suspension for Above Knee Amputees
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stony Brook University (Other)
Collaborators: Otto Bock Healthcare Products GmbH (Industry)
Responsible Party: Principal Investigator, Eric Lamberg, Clinical Associate Professor, Stony Brook University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 197622
Record Dates: First submitted 2011-08-16; First posted 2012-03-21 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Amputation
Keywords: Lower limb loss; Leg amputation; walking study; socket technology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Socket wall height (Experimental)
  Interventions: Device: Vacuum assisted socket technology (Harmony System, Otto Bock Healthcare)

INTERVENTIONS:
Device: Vacuum assisted socket technology (Harmony System, Otto Bock Healthcare) — The brim height of the socket will be systematically reduced

SUMMARY:
Individuals with transfemoral (TF) amputation (above the knee amputation) may benefit from a socket that uses vacuum assisted suspension (VAS) to hold the socket onto the amputated limb. VAS may improve stability, weight bearing, comfort, proprioception, limb health, and function. To date, there is no evidence to support whether VAS alters balance, kinematics, and kinetics when walking for TF amputees as compared to conventional socket suspension technology. Further, there is question regarding what the optimal height of the socket should be to maintain stability and function. So long as stability is not sacrificed, it may be advantageous to lower the height of the socket to allow full hip motion and improve sitting comfort. The purpose of this investigation is to assess if the socket height alters the motion of the leg and changes the way one walks when using VAS compared to conventional socket suspension technology. In this study, TF amputees will be fitted with a VAS socket that will be attached to their current prosthesis using similar alignment. Individuals will be assessed while walking on a level floor and during stair negotiation while wearing the prosthesis with the VAS socket at various socket heights as well as their current socket. Additionally, balance and socket standing and sitting comfort will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 21 and 75 with a transfemoral amputation.
* Limited household ambulators (K1) to those considered unlimited community ambulators (K4).
* People who are comfortably fitted with a prosthesis for at least 6 months.

Exclusion Criteria:

* People with severe cardiac or pulmonary disease that limits ability to walk.
* People with too much discomfort and/or pain.
* People with active wounds on their residual limb or other foot.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Gait changes | 1 day
  Step length, stride length, stance time, swing time, velocity

SECONDARY OUTCOMES:
Comfort | 1 day
Balance | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Eric M Lamberg, EdD, PT, Principal Investigator — Stony Brook University
Locations (2):
- United States (2):
  - Stony Brook University, Stony Brook, New York
  - Long Island Orthotics and Prosthetics, West Babylon, New York